CLINICAL TRIAL: NCT03333057
Title: A Phase 2, Multi-Center, Randomized, Double-Masked, Saline-Controlled Study to Evaluate the Effect of Perfluorohexyloctane (NOV03) at Two Different Dosing Regimens on Signs and Symptoms of Dry Eye Disease (DED)
Brief Title: Perfluorohexyloctane (NOV03) for the Treatment of Signs and Symptoms of Dry Eye Disease (DED)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novaliq GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NVU-002 (SEECASE)
Record Dates: First submitted 2017-11-02; First posted 2017-11-06 (Actual); Results first posted 2021-05-24 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2019-10

CONDITIONS: Dry Eye Disease (DED)
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- NOV03 4 times daily (QID) (Experimental): Perfluorohexyloctance solution 4 times daily (QID)
  Interventions: Drug: NOV03
- NOV03 2 times daily (BID) (Experimental): Perfluorohexyloctance solution 2 times daily (BID)
  Interventions: Drug: NOV03
- Placebo 4 times daily (QID) (Placebo Comparator): Saline solution (0.9% sodium chloride solution) 4 times daily (QID)
  Interventions: Drug: Placebo
- Placebo 2 times daily (BID) (Placebo Comparator): Saline solution (0.9% sodium chloride solution) 2 times daily (BID)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: NOV03 — Perfluorohexyloctane
  Arms: NOV03 2 times daily (BID); NOV03 4 times daily (QID)
Drug: Placebo — Saline solution (0.9% sodium chloride solution)
  Arms: Placebo 2 times daily (BID); Placebo 4 times daily (QID)

SUMMARY:
This study will evaluate the efficacy, safety and tolerability of perfluorohexyloctane (NOV03) at two different dosing regimens compared to saline solution in subjects with Dry Eye Disease (DED).

ELIGIBILITY:
Inclusion Criteria:

* Signed ICF (Informed Consent Form)
* Subject-reported history of Drye Eye Disease (DED) in both eyes
* Ability and willingness to follow instructions, including participation in all study assessments and visits

Exclusion Criteria:

* Women who are pregnant, nursing or planning pregnancy
* Unwillingness to submit a blood pregnancy test at screening and the last visit (or early termination visit) if of childbearing potential, or unwillingness to use acceptable means of birth control
* Clinically significant slit-lamp findings or abnormal lid anatomy at screening
* Ocular/peri-ocular malignancy
* History of herpetic keratitis
* Active ocular allergies or ocular allergies that are expected to be active during the study
* Ongoing ocular or systemic infection
* Wear contact lenses within 1 month prior to screening or anticipated use of contact lenses during the study
* Intra-ocular surgery or ocular laser surgery within the previous 6 months, or have planned ocular and/or lid surgeries over the study period
* Presence of uncontrolled systemic diseases
* Presence of known allergy and/or sensitivity to the study drug or saline components
* Use of any topical steroids treatments, topical cyclosporine, lifitegrast, serum tears or topical anti-glaucoma medication within 2 months prior to screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Actual)
Dates: Start 2018-01-03 (Actual); Primary Completion 2018-05-18 (Actual); Study Completion 2018-07-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonja Kroesser, PhD, Study Director — Novaliq GmbH
Locations (9):
- United States (9):
  - Investigational site, Artesia, California
  - Investigational Site, Newport Beach, California
  - Investigational Site, Santa Ana, California
  - Investigational Site, Torrance, California
  - Investigational site, Jacksonville, Florida
  - Investigational Site, Lake Villa, Illinois
  - Investigational Site, Kansas City, Missouri
  - Investigational Site, Pennington, New Jersey
  - Investigational Site, Nashville, Tennessee

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Tauber J, Wirta DL, Sall K, Majmudar PA, Willen D, Krosser S; SEECASE study group. A Randomized Clinical Study (SEECASE) to Assess Efficacy, Safety, and Tolerability of NOV03 for Treatment of Dry Eye Disease. Cornea. 2021 Sep 1;40(9):1132-1140. doi: 10.1097/ICO.0000000000002622. PMID 33369937
- See also: Publication of Study Results in Cornea — https://pubmed.ncbi.nlm.nih.gov/33369937/

RESULTS

PARTICIPANT FLOW:
Groups:
- NOV03 4 Times Daily (QID): Perfluorohexyloctance solution 4 times daily
  NOV03: Perfluorohexyloctane
- Placebo BID/QID: Saline solution (0.9% sodium chloride solution) 2/4 times daily (BID/QID)
  Placebo: Saline solution (0.9% sodium chloride solution)
Period: Overall Study
Arm/Group | NOV03 2 Times Daily (BID) | NOV03 4 Times Daily (QID) | Placebo BID/QID
Started | 111 | 114 | 111
Completed | 105 | 110 | 108
Not Completed | 6 | 4 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | NOV03 2 Times Daily (BID) | NOV03 4 Times Daily (QID) | Placebo BID/QID | Total
Number analyzed (Participants) | 111 | 114 | 111 | 336
Age, Continuous [Mean (Full Range); unit: years] | 54.0 [22 to 86] | 53.0 [22 to 86] | 53.8 [19 to 85] | 53.6 [19 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84 | 79 | 80 | 243
  Male | 27 | 35 | 31 | 93
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 30 | 21 | 77
  Not Hispanic or Latino | 85 | 84 | 90 | 259
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 20 | 18 | 21 | 59
  Native Hawaiian or Other Pacific Islander | 0 | 2 | 0 | 2
  Black or African American | 13 | 13 | 8 | 34
  White | 78 | 80 | 81 | 239
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 111 | 114 | 111 | 336

OUTCOME MEASURES:

1. Primary Outcome: Corneal Fluorescein Staining (CFS) Total (National Eye Institute (NEI) Grading)
Description: The primary efficacy variable was comparison of absolute and change from baseline between treatments for total Corneal Fluorescein Staining (tCFS) according to the National Eye Institute grading (NEI Scale) at week 8
  The NEI Scale is a standardized grading system. 0-3 is used for each of the five areas on each cornea. Grade 0 will be specified when no staining is present. The maximum total score for each eye is 15. Higher values describe greater staining and corneal damage.
Time Frame: baseline and 2 months
Measure: Mean (95% Confidence Interval); unit: score on a scale
Groups:
- NOV03 4 Times Daily (QID): Perfluorohexyloctance solution 4 times daily
  NOV03:Perfluorohexyloctane
Arm/Group | NOV03 2 Times Daily (BID) | NOV03 4 Times Daily (QID) | Placebo BID/QID
Number analyzed (Participants) | 111 | 114 | 111
score on a scale | -1.78 [-2.27 to -1.30] | -2.11 [-2.59 to -1.63] | -0.93 [-1.41 to -0.45]

ADVERSE EVENTS:
Time Frame: whole study duration (8 weeks per patient)
Arm/Group | NOV03 2 Times Daily (BID) | NOV03 4 Times Daily (QID) | Placebo BID/QID
All-Cause Mortality (participants affected / at risk) | 0/111 | 0/114 | 0/111
Serious Adverse Events (participants affected / at risk) | 1/111 | 3/114 | 0/111
Other Adverse Events (participants affected / at risk) | 1/111 | 4/114 | 3/111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOV03 2 Times Daily (BID) (N=111) | NOV03 4 Times Daily (QID) (N=114) | Placebo BID/QID (N=111)
Diverticulum (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NOV03 2 Times Daily (BID) (N=111) | NOV03 4 Times Daily (QID) (N=114) | Placebo BID/QID (N=111)
Vision blurred (Eye disorders) | 0 (0) | 2 (2) | 1 (1)
Instillation site pain (General disorders) | 1 (2) | 2 (2) | 0 (0)
Instillation site irritation (General disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-12-07): https://cdn.clinicaltrials.gov/large-docs/57/NCT03333057/Prot_SAP_000.pdf